CLINICAL TRIAL: NCT06336161
Title: Comparison Between Ultrasound-Guided Erector Spinae Plane Block Versus Ultrasound-Guided Caudal Injection in Lumbosacral Spine Surgeries for Postoperative Pain Management
Brief Title: Comparison Between Ultrasound-Guided Erector Spinae Plane Block Versus Ultrasound-Guided Caudal Injection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Khalil Elsayed Khalil, Cairo,Egypt, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESPB versus CEI
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A ( Erector Spinae Plane Block) (Active Comparator): About 40 patients who will be subjected to Ultrasound-Guided Erector Spinae Plane Block.for Postoperative Pain Management
  Interventions: Drug: Fentanyl
- Group B (Caudal Injection) (Active Comparator): About 40 patients who will be subjected to Ultrasound-Guided Caudal Injection in Lumbosacral Spine Surgeries for Postoperative Pain Management
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — to compare between Ultrasound-Guided ESPB and Ultrasound-Guided CEI for postoperative pain relief in patients who underwent lumbosacral surgeries.
  Other Names: propofol 2Mg/Kg

SUMMARY:
Patient-controlled analgesia is typically used to relieve postoperative pain. Patient-controlled analgesia, on the other hand, is prone to opioid-related side effects. Furthermore, standard postoperative analgesia has a limited analgesic impact. If postoperative lumbosacral spine pain is not successfully treated, it can progress to chronic pain, compromising patients' quality of life.

The methods of access for epidural injections are characterized as transforaminal, interlaminar, or caudal. Caudal epidural injections (CEI) are often utilized as a diagnostic or therapeutic tool in a range of lumbosacral-originating spinal pain problems, and they are especially useful in patients with complicated lumbar epidural access diseases, such as post laminectomy syndrome. It is regarded as a very simple treatment in the realm of interventional pain management, and it is also recognized to have a reduced risk of inadvertent Dural puncture than other epidural techniques

DETAILED DESCRIPTION:
Patient-controlled analgesia is typically used to relieve postoperative pain. Patient-controlled analgesia, on the other hand, is prone to opioid-related side effects. Furthermore, standard postoperative analgesia has a limited analgesic impact. If postoperative lumbosacral spine pain is not successfully treated, it can progress to chronic pain, compromising patients' quality of life.

Major lumbosacral surgery results in considerable postoperative discomfort that normally lasts at least three days. According to several research, the most discomfort occurs in the first four postoperative hours and gradually decreases by the third postoperative day. Efficient and safe postoperative analgesic treatments following lumbosacral surgery are useful for early recovery and hence required.

Traditional caudal epidural injections, on the other hand, pose a potential risk of epidural venous plexus or dura penetration, with the incidence of accidental intravascular injections, as confirmed by contrast enhanced fluoroscopy, ranging from 11 to 42% in patients who had received caudal epidural injections. Furthermore, there have been a few instances of unintended Dural puncture during the caudal approach because of an unusually low Dural sac termination in the sacral canal.

Such complications of intravascular and intrathecal drug injections might result in systemic toxicity of local anesthetics and complete spinal anesthesia. Thus, ultrasonography (US) can be utilized to guide caudal injections, increasing the efficacy of pain treatment while decreasing the risk of complications and incorrect injections. Previous investigations shown the feasibility of using ultrasound to locate the sacral hiatus and guide the needle into the caudal epidural area, with a reported success rate of 100%.

Another technique for postoperative pain relief is the Erector spinae plane block (ESPB), which was introduced in 2016. It is a relatively new regional anesthesia technique in which local anesthetic is injected into the fascial plane between the transverse process of the vertebra and the erector spinae muscles. It has acquired favor in perioperative analgesia for a variety of surgical procedures, including breast, thoracic, abdominal, and lumbar spine operations.

The addition of US to ESPB allows the needle to be guided to efficiently deposit the anesthetic agents deep to the erector spinae muscle, resulting in the blockage of the ventral and dorsal rami of many spinal neurons, boosting the efficiency of pain control.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lumbosacral spine surgeries from (L4-L5) level to end of spinal cord.
* American society of anesthesiologists' classification (ASA) I & II.

Exclusion Criteria:

* Patient's refusal.
* History of any previous back surgeries.
* History of any spinal cord deformities e.g., Scoliosis, Lordosis, Kyphosis, Ankylosing Spondylitis
* Bleeding disorders (platelets count < 80,000; International normalized ratio >1.4; PC< 70%) and coagulopathies.
* Skin lesion, wounds, or infection at the injection site.
* Known allergy to local anesthetic drugs.
* Peripheral and Central Neuropathy.
* Patients with pre-operative opioid consumption.
* Chronic opioids or analgesics users.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of Post-operative Pain | the first 24 hours postoperatively
  Assessment of Pain after operations will be evaluated using the VAS consisting of a horizontal or vertical line, 10 centimeters long (100 mm) anchored at the extremes by two verbal descriptors referring to the pain status

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Monir, Professor, Study Chair — Anesthesiology, Intensive care, and Pain Management, Faculty of Medicine, Al-Azhar University
Locations (1):
- Al-Azhar University hospitals, Cairo, Egypt

REFERENCES:
- [Result] Patel Y, Ramachandran K, Shetty AP, Chelliah S, Subramanian B, Kanna RM, Shanmuganathan R. Comparison Between Relative Efficacy of Erector Spinae Plane Block and Caudal Epidural Block for Postoperative Analgesia in Lumbar Fusion Surgery- A Prospective Randomized Controlled Study. Global Spine J. 2025 Mar;15(2):639-647. doi: 10.1177/21925682231203653. Epub 2023 Sep 22. PMID 37737097
- [Result] Shah M, Halalmeh DR, Sandio A, Tubbs RS, Moisi MD. Anatomical Variations That Can Lead to Spine Surgery at the Wrong Level: Part III Lumbosacral Spine. Cureus. 2020 Jul 28;12(7):e9433. doi: 10.7759/cureus.9433. PMID 32864257
- See also: Acute Postoperative Pain: Patient-Controlled Analgesia — https://link.springer.com/chapter/10.1007/978-3-030-87266-3_3
- See also: Caudal epidural steroid injection ultrasound-guided versus fluoroscopy-guided in treatment of refractory lumbar disc prolapse with radiculopathy — https://ejrnm.springeropen.com/articles/10.1186/s43055-020-00388-8